CLINICAL TRIAL: NCT06838169
Title: Effects of Breathıng Exercıses wıth Vırtual Realıty Glasses on Anxıety Levels, Sleep Qualıty and Respıratory Parameters in Heart Faılure Patıents
Brief Title: The Effect of Vırtual Realıty Glasses on Heart Faılure Patıents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bayburt University (Other)
Responsible Party: Principal Investigator, Servet KALYONCUO, Research Assistant, Bayburt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RCS2253148
Record Dates: First submitted 2025-01-16; First posted 2025-02-20 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure
Keywords: Heart failure; Virtual reality glasses; Anxiety; Respiration; Sleep Quality
MeSH Terms: conditions — Heart Failure; Anxiety Disorders; Respiratory Aspiration; Sleep Initiation and Maintenance Disorders | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality glasses + breathing exercise app (Experimental): Virtual reality glasses + breathing exercise app
  Interventions: Behavioral: Virtual reality glasses; Behavioral: breathing exercise
- Breathing exercise practice (Active Comparator): Breathing exercise practice
  Interventions: Behavioral: breathing exercise
- Kontrol (No Intervention): No application will be made

INTERVENTIONS:
Behavioral: Virtual reality glasses — virtual reality glasses application
  Arms: Virtual reality glasses + breathing exercise app
Behavioral: breathing exercise — breathing exercise app
  Arms: Breathing exercise practice; Virtual reality glasses + breathing exercise app

SUMMARY:
Anxiety and sleep disorders are among the most common symptoms in heart failure patients. In addition to pharmacological methods for anxiety and sleep disorders, non-pharmacological methods can also be used. Among these, anxiety and sleep disorders can be prevented with virtual reality glasses aimed at distraction. This study will be conducted to evaluate the effect of breathing exercises performed with virtual reality glasses on anxiety, sleep quality, and respiratory parameters. The study will be conducted with a total of 45 patients, 15 virtual reality glasses + breathing exercises, 15 breathing exercises, and 15 controls. Those in the virtual reality glasses + breathing exercises group will perform breathing exercises with virtual reality glasses once a day for 7 days. Those in the breathing exercises group will perform only breathing exercises once a day for 7 days. Anxiety, sleep disorders, and respiratory parameters of the patients will be examined.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Verbal communication,
* Place and time oriented,
* Without any psychiatric illness,
* Patients diagnosed with HF with NYHA class III-IV symptoms,
* Left ventricular ejection fraction ≥50% (LVEF-CF/HFpEF), between 40-49% (SEF-CF/HFmrEF), HF below 40% (DEF-CF/HFrEF),
* High levels of natriuretic peptides (BNP>35 pg/mL and/or NTproBNP>125 pg/mL),
* There is no deformity or diagnosis related to the musculoskeletal system that may prevent breathing exercise,
* Chronic diseases such as hypertension (Stage 1 and 2 HT) and diabetes mellitus are stable and the treatment for these diagnoses has not been changed in the last month,
* Who have not previously received respiratory exercise training and have not participated in a rehabilitation program,
* Patients who volunteer to participate in the study will be included in the study

Exclusion Criteria:

* Life signs are so abnormal as to preclude intervention,
* Patients with migraine, vertigo, active nausea-vomiting, headache, dizziness will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety level | Apply the morning before application and the morning 7 days after application.
  Turkish adaptation of the state-trait anxiety inventory short version (STAIS-5, STAIT-5). This form is a 4-point Likert type. It is an easy-to-apply inventory consisting of a total of 10 statements. As the score obtained in this form increases, the level of anxiety also increases.

SECONDARY OUTCOMES:
Sleep Quality | Apply the morning before application and the morning 7 days after application.
  Richard Campbell Sleep Quality Scale (RCSQ) for sleep quality level assessment.This form is a 6-item scale. According to the scale scoring, a score between "0-25" indicates very poor sleep, and a score between "76-100" indicates very good sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Servet Kalyoncuo, Principal Investigator — ERCİYES UNIVERSITY
Locations (1):
- T.C. Erciyes University Faculty of Medicine Hospitals, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polikandrioti M, Goudevenos J, Michalis LK, Koutelekos J, Kyristi H, Tzialas D, Elisaf M. Factors associated with depression and anxiety of hospitalized patients with heart failure. Hellenic J Cardiol. 2015 Jan-Feb;56(1):26-35. PMID 25701969
- See also: referances — https://pubmed.ncbi.nlm.nih.gov/25701969/